CLINICAL TRIAL: NCT06536504
Title: A Randomized Controlled Trial to Assess the Impact of Live and Recorded Music-Based Interventions on Pre-operative Stress, Mood, Pain and Biomarkers, in Neurosurgical Patients (Music-STAR Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0082; NCI-2024-06549 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stress; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients: Simulated Live Music (Experimental): Patients will be screened for eligibility, enrolled in the study and randomized 1:1:1.
  Interventions: Other: Steinway Spirio M recording/player piano
- Patients: Recorded Music (Experimental): Patients will be screened for eligibility, enrolled in the study and randomized 1:1:1.
  Interventions: Other: Steinway Spirio M recording/player piano
- Patients: Control: No Music (Experimental): Patients will be screened for eligibility, enrolled in the study and randomized 1:1:1.
  Interventions: Other: Steinway Spirio M recording/player piano

INTERVENTIONS:
Other: Steinway Spirio M recording/player piano — Patients will be equally randomized into one of the three arms (simulated live music, recorded music, or no music) applying the random permutated block. Randomization will be conducted via an approved institutional database with the randomization list generated by the study statistician.

SUMMARY:
The study plans to enroll a total of 132 patients. The goal of this study is to measure pre-and post-music intervention changes in patients' vital signs, serum- and plasma-level biomarkers by broad-spectrum proteomics analysis, metabolic analysis, and perceived pain, anxiety, and mood states as measured by validated questionnaires (STAI-S, POMS-SF, and VASP). We will collect demographic information on each participant. Participants will also complete the Brief Musical Experience Questionnaire (BMEQ) to investigate potential links between susceptibility to music-induced anxiolysis and prior musical training, preference and exposure.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the effects of the two (live and recorded) prescribed preoperative containing CER on physiologic and perceived stress in patients undergoing Neurosurgery.
* To evaluate the effects of those two music interventions on serum- and plasma-level stress biomarkers and cytokines in those patients.

Secondary Objectives:

• To measure correlative effects of demographic variables, prior musical training, experience, preference, and exposure to music.

ELIGIBILITY:
Inclusion Criteria

1) Patients undergoing neurosurgical procedures will be eligible to enroll in this study.

Exclusion Criteria

1. Patient is unable or unwilling to provide informed consent.
2. Patient is deaf or hearing-disabled.
3. Patient is less than 18 years in age.
4. Patient was previously enrolled in the study.
5. Non-English-speaking patients (patient must be fluent in English and not require translation services per MDACC institutional policy.
6. Subjects on contact isolation precautions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Stress and mood changes | Through study cmpletion
  Pre-post intervention changes in physiologic and perceived stress and mood changes by BP, STAI-S, VASP and POM-S.
Stress biomarkers | Through study completion
  Proteomic and metabolomic analyses, in stress biomarkers and cytokines including IL-6, cortisol and epinephrine.

SECONDARY OUTCOMES:
BMEQ (Brief Music Experience Questionnaire) | Through study completion
  Approximately 15 minutes to complete each time)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Rui, DMA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org